CLINICAL TRIAL: NCT02531724
Title: Effects of Levosimendan in Acute Kidney Injury After Cardiac Surgery
Acronym: LEVOAKI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lukas Lannemyr, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SahlgrenskaUHThoraxLL3
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Acute Kidney Injury; Renal Insufficiency, Acute
Keywords: acute kidney injury; cardiac surgery; renal blood flow; levosimendan
MeSH Terms: conditions — Acute Kidney Injury | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levosimendan (Active Comparator): Levosimendan will be given as a loading dose of 12 ug/kg during 30 minutes, and then a continuous infusion of 0,1 ug/kg/min for 180 minutes.
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): Sodium chloride will be given as a loading dose during 30 minutes and then a continuous infusion for 180 minutes at a rate mimicking the levosimendan group above.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan
  Other Names: Simdax
  Arms: Levosimendan
Drug: Placebo — Sodium chloride
  Arms: Placebo

SUMMARY:
Acute kidney injury (AKI) is a common complication after cardiac surgery. Mismatch in renal oxygen demand-supply may be an important pathogenetic factor. Levosimendan has been shown to improve renal blood flow, glomerular filtration rate and renal oxygenation in healthy controls after cardiac surgery.

In order to investigate the effect of levosimendan in patients with AKI after cardiac surgery, the investigators plan a randomized placebo controlled trial. 30 patients will receive levosimendan or placebo. Renal blood flow and filtration fraction will be measured using infusion clearance technique of para-aminohippuric acid and Chromium ethylenediaminetetraacetic acid (Cr-EDTA) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the cardiothoracic intensive care after cardiac surgery with cardiopulmonary bypass
* Acute kidney injury, defined as increase in S-creatinine 50% or 27 mol/L
* Normal S-creatinine before surgery

Exclusion Criteria:

* Ongoing treatment with inotropic drugs (not norepinephrine)
* Central venous oxygen saturation (ScvO2) < 60% despite optimization of hematocrit and volume status
* Need of renal replacement therapy
* Ongoing bleeding
* Patient or next of kin does not consent with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Renal blood flow | 5 Hours
  Renal blood flow will be measured using infusion clearance technique of para-aminohippuric acid. Measurements will be made in duplicates before and after administration of the study drug.
Glomerular filtration rate | 5 Hours
  Filtration fraction will be determined using be measured using infusion clearance technique of Chromium ethylenediaminetetraacetic acid (Cr-EDTA). Measurements will be made in duplicates before and after administration of the study drug. Glomerular filtration rate will be calculated as the filtration fraction multiplied by renal plasma flow.

SECONDARY OUTCOMES:
Serum creatinine | 4 days
  Measurement of serum creatinine will be made daily the first 4 days after the study

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Professor, Study Director — Sahlgrenska Academy, dept of clinical science
Locations (1):
- Department of thoracic anesthesia, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Bragadottir G, Redfors B, Ricksten SE. Effects of levosimendan on glomerular filtration rate, renal blood flow, and renal oxygenation after cardiac surgery with cardiopulmonary bypass: a randomized placebo-controlled study. Crit Care Med. 2013 Oct;41(10):2328-35. doi: 10.1097/CCM.0b013e31828e946a. PMID 23921271
- [Derived] Tholen M, Ricksten SE, Lannemyr L. Effects of levosimendan on renal blood flow and glomerular filtration in patients with acute kidney injury after cardiac surgery: a double blind, randomized placebo-controlled study. Crit Care. 2021 Jun 12;25(1):207. doi: 10.1186/s13054-021-03628-z. PMID 34118980